CLINICAL TRIAL: NCT01279317
Title: The Effect of Vinegar Co-ingestion on Postprandial Glucose Control in Type 2 Diabetes Patients
Brief Title: Vinegar Co-ingestion in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MEC 10-3-035
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Results first posted 2011-10-03 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acetic Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- vinegar co-ingestion (Experimental): 25 ml vinegar is added to glucose containing beverage
  Interventions: Dietary Supplement: vinegar co-ingestion
- Placebo co-ingestion (Placebo Comparator): 25 ml vinegar is substituted by 25 ml water
  Interventions: Dietary Supplement: placebo co-ingestion

INTERVENTIONS:
Dietary Supplement: placebo co-ingestion — 25 ml water co-ingested with a glucose-containing beverage
  Arms: Placebo co-ingestion
Dietary Supplement: vinegar co-ingestion — 25 ml vinegar (1 g acetic acid) co-ingested with a glucose-containing beverage
  Other Names: vinegar; acetic acid
  Arms: vinegar co-ingestion

SUMMARY:
The main objective of this study is to assess the acute effect of co-ingested vinegar on postprandial plasma glucose levels in type 2 diabetes patients.

DETAILED DESCRIPTION:
Plasma glucose and insulin concentrations are assessed over the 2 hr period following ingestion of carbohydrate-rich beverage with or without added vinegar.

ELIGIBILITY:
Inclusion Criteria:

* male type 2 diabetes
* overweight or obese
* 40-70 yrs

Exclusion Criteria:

* incident cardiovascular events during last year
* peptic ulcer, duodenal ulcer, oesophageal reflux
* antacids, H2 receptor blocker, proton pump inhibitors, NSAIDS, prokinetic agents

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment by advertisements in local newspaper
Pre-assignment Details: none applicable
Groups:
- Vinegar Co-ingestion First, Then Placebo Co-intestion: First acute experiment with vinegar-coingestion (1 day), after 1 week washout, experiment with placebo co-ingestion (1 day).
- Placebo Co-ingestion First, Then Vinegar Co-ingestion: First acute experiment with placebo-coingestion (1 day), after 1 week washout experiment with vinegar co-ingestion (1 day).
Period: Period 1
Arm/Group | Vinegar Co-ingestion First, Then Placebo Co-intestion | Placebo Co-ingestion First, Then Vinegar Co-ingestion
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Washout
Arm/Group | Vinegar Co-ingestion First, Then Placebo Co-intestion | Placebo Co-ingestion First, Then Vinegar Co-ingestion
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Vinegar Co-ingestion First, Then Placebo Co-intestion | Placebo Co-ingestion First, Then Vinegar Co-ingestion
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Vinegar Co-ingestion: All participants performed both intervention periods.
Arm/Group | Vinegar Co-ingestion
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 65 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Region of Enrollment [Number; unit: participants]
  Netherlands | 12

OUTCOME MEASURES:

1. Primary Outcome: Postprandial Glycemic Incremental Area Under the Curve
Description: area under the plasma glucose concentration curve, above the baseline plasma glucose, measured over 2 hr following ingestion of a the intervention beverages
Time Frame: 2 hr
Population: all subjects completed study and are included in analysis
Measure: Mean (Standard Error); unit: mmol/L / 2hr
Arm/Group | Vinegar Co-ingestion | Placebo Co-ingestion
Number analyzed (Participants) | 12 | 12
mmol/L / 2hr | 739 (74) | 759 (75)

ADVERSE EVENTS:
Arm/Group | Vinegar Co-ingestion
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No